CLINICAL TRIAL: NCT05676359
Title: Knowledge of Living Will in Patients With Rheumatic Diseases. A Case-control Study
Brief Title: Knowledge of Living Will in Patients With Rheumatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Virginia Pascual Ramos, Principal Investigator, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Other Study IDs: IRE-4312
Record Dates: First submitted 2022-12-15; First posted 2023-01-09 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Rheumatic Disorder
Keywords: Rheumatic diseases; living will
MeSH Terms: conditions — Rheumatic Diseases | interventions — ametantrone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with rheumatic diseases from the outpatient clinic at a tertiary care level in Mexico City
  Interventions: Other: Health Assessment Questionnaire (HAQ); Other: Depression, Anxiety and Stress Scale (DASS-21); Other: Brief Resilient Coping Scale; Other: WHOQOL-BREF; Other: Routine assessment of patient index data 3 (RAPID-3); Other: Rheumatic disease comorbidity index; Other: Living will questionnaire; Other: Perceptions of Health Outcomes Questionnaire
- Controls: Two patients´ relatives of the same sex, age ± five years and who are known to be healthy
  Interventions: Other: Health Assessment Questionnaire (HAQ); Other: Depression, Anxiety and Stress Scale (DASS-21); Other: Brief Resilient Coping Scale; Other: WHOQOL-BREF; Other: Rheumatic disease comorbidity index; Other: Living will questionnaire; Other: Perceptions of Health Outcomes Questionnaire

INTERVENTIONS:
Other: Health Assessment Questionnaire (HAQ) — The HAQ is based on five patient-centered dimensions: disability, pain, medication effects, costs of care, and mortality
Other: Depression, Anxiety and Stress Scale (DASS-21) — DASS-21 is a set of three self-report scales designed to measure the emotional states of depression, anxiety, and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content
Other: Brief Resilient Coping Scale — Brief Resilient Coping Scale is a 4-item measure designed to capture tendencies to cope with stress in a highly adaptive manner
Other: WHOQOL-BREF — WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health, psychological health, social relationships, and environmental health; it also contains QOL and general health items
Other: Routine assessment of patient index data 3 (RAPID-3) — RAPID- 3 measures: function, pain, and patient global estimate of status. Each of the 3 individual measures is scored 0 to 10, for a total of 30
  Groups: Cases
Other: Rheumatic disease comorbidity index — It is rated from 0 to 9 and comprises 11 comorbid conditions including lung disease, cardio-vascular disease, hypertension, diabetes, fracture, depression, cancer, and gastrointestinal ulcer
Other: Living will questionnaire — A questionnaire with 17 items about knowledge of the living will.
Other: Perceptions of Health Outcomes Questionnaire — A questionnaire with 7 items about the probability of quitting the job, getting an infectious disease, requiring emergency medical attention, hospitalization or intensive care, dependence and death.

SUMMARY:
The living will is a legal document derived from a communication and deliberation process, medical ethical aspect, currently regulated in Mexico by the General Health Law and the Health Law of Mexico City.

Knowledge of living will in the population with chronic diseases, including rheumatic diseases, has been little addressed. Most patients do not know what the living will document is, so they do not carry it out and others, despite knowing it, have a passive attitude toward doing it.

DETAILED DESCRIPTION:
A study will be carried out on patients with rheumatic diseases and healthy family controls. Patients will be selected from those attending the Department of Immunology and Rheumatology in Mexico City outpatient department, including consecutive cases.

The patients will be assessed for their quality of life and disability. Patients and controls will be evaluated on the knowledge of living will, their perceptions about specific health outcomes, sociodemographic characteristics, comorbidities, and psychiatric pathology.

ELIGIBILITY:
Inclusion Criteria:

Cases

* Patients with a rheumatic disease diagnostic by a rheumatologist
* Patients with rheumatic diseases attending the Department of Immunology and Rheumatology in Mexico City outpatient department
* Patients who agree to participate in the study, who complete and sign the informed consent Controls
* Relative of a patient with rheumatic diseases of the same sex and age ± 5 years, without known rheumatic and/or chronic disease and without the use of pharmacological treatment for more than 7 days during the month before study entry.

Exclusion Criteria:

Cases

* Patients with severe diseases or in palliative care by a rheumatologist

Controls

- Withdrawal of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from those attending the Department of Immunology and Rheumatology in Mexico City outpatient department, and the controls will be patients´ relatives of the same sex, age ± five years and who are known to be healthy
Sampling Method: Non-Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge of the living will with the living will questionnaire (locally development) | 1 day At study inclusion (After their rheumatology consultation)
  To evaluate the knowledge of the living will, using the living will questionnaire (locally development), among the patients with rheumatic diseases and healthy controls.
Perceptions of Health Outcomes with the perceptions of health outcomes questionnaire (locally development) | 1 day At study inclusion (After their rheumatology consultation)
  To evaluate the perceptions of the of health outcomes using the perceptions of health outcomes questionnaire (locally development), among the patients with rheumatic diseases and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Pascual-Ramos, Dr., Principal Investigator — National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No